CLINICAL TRIAL: NCT06955403
Title: How Does PRECISION7® for Astigmatism Perform in Current and Successful Acuvue® Oasys for Astigmatism Wearers?
Brief Title: Acuvue Oaysis Contact Lens Wearers Being Refit Into P7 Contact Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Collaborators: Eminent Ophthalmic Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P7
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Contact Lens Comfort

STUDY DESIGN:
Intervention Model Description: This will be a prospective study to understand if satisfied AOA CL wearers can be successfully refit into P7A CLs. The Primary Endpoint will be analyzed as the proportion of participants who have CLDEQ-8 scores <12 at the end of the study; thus, no comparison will occur with the Primary Endpoint and no formal sample size calculation can be performed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PRECISION7 (Experimental): Determine the likelihood of successfully refitting a satisfied Acuvue Oaysis Contact Lens wearers into P7A CLs.
  Interventions: Device: Precision 7 contact lenses

INTERVENTIONS:
Device: Precision 7 contact lenses — Acuvue Oaysis contact lens wearers have will be refit into precision 7 contact lenses.

SUMMARY:
Determine the likelihood of successfully refitting a satisfied AOA CL wearers into P7A CLs

DETAILED DESCRIPTION:
PRECISION7m for Astigmatism is a 1-week, silicone hydrogel (serafilcon A), daily wear, contact lens (CL) with extended wear approval made of a novel material that incorporates the Activ-Flo System. The Activ-Flo System has a moisturizing agent within the CL matrix, which allows for continual release of the moisturizing agents while also providing up to 16 hours of comfortable wear and precise vision for the life of the CL. While initial P7A data are promising, the literature currently lacks a targeted study aimed at determining how patients perform in P7A after transitioning out of other commonly prescribed silicone hydrogel CLs. This transition could be particularly important for patients who have astigmatism given that they tend to struggle with CLs more than spherical CL wearers.1 Thus, the purpose of this study is to determine the success rate of refitting current, satisfied ACUVUE OASYS for Astigmatism CL wearers into P7A. Understanding how a P7A CL wearer reacts to transitioning into P7A from AOA will provide valuable information to partitioners for patient educational purposes, and it will provide credence for refitting successful AOA patients into the newer P7A technology, which could help grow the P7A CL market by not limiting P7A refits to problem-solving events.

ELIGIBILITY:
• Inclusion Criteria: Adults, 18- to 40-year-old, AOA CL wearers with best-corrected 20/20 visual acuity or better.

* Participants will be required to have worn AOA CLs for at least 3 months in the past year and currently wearing these CLs.
* All participants will be required to have a CLDEQ-8 score <12 while wearing their habitual CLs (AOA CLs) and to indicate that they are satisfied with AOA CLs (Yes/No).
* Participants will be required to be able to wear P7A CLs (astigmatism ≥0.75D OD/OS).
* Astigmatism ranging from 0.75 D to 2.50 D in each eye
* Participants will be required to wear the study CLs for ≥13 hours with no overnight wear
* Participants will be willing to wear the CL every day of the week, except during the washout period
* Participants will be required to provide a glasses prescription that is less than 3 years old
* -
* Exclusion Criteria:
* - Have presbyopia and/or need a reading add as determined during their initial manifest refraction
* Have worn P7A in the past
* Are past rigid CL wearers
* Have a history of being diagnosed with dry eye or ocular allergies
* Have known systemic health conditions that are thought to alter tear film physiology
* Have a history of viral eye disease
* Have a history of ocular surgery
* Have a history of severe ocular trauma
* Have a history of corneal dystrophies or degenerations
* Have active ocular infection or inflammation
* Are currently using isotretinoin-derivatives or ocular medications
* Are pregnant or breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Likert questionnaire | 1 week
  1. Likelihood of continuing to wear P7A, 2. Overall satisfaction while wearing P7A, 3. Overall vision while wearing P7A, 4. End of day comfort while wearing P7A, 5. End of day vision while wearing P7A, 6. Overall comfort while wearing P7A, 7. Ability to play sports and perform fitness actives while wearing P7A, 8. Ability to use digital devices while wearing P7A (questions attached). 9. Would recommend the study CLs to a friend.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Lievens, Principal Investigator — The Southern College of Optometry
Locations (1):
- The Southern College of Optometry, Memphis, Tennessee, United States